CLINICAL TRIAL: NCT01288794
Title: The Use of Human Albumin for the Treatment of Ascites in Patients With Hepatic Cirrhosis: a Multicenter, Open-label Randomized Clinical Trial
Brief Title: Human Albumin for the Treatment of Ascites in Patients With Hepatic Cirrhosis
Acronym: ANSWER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Mauro Bernardi, Full Professor of Medicine, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FARM6P824B; 2008-000625-19 (EudraCT Number)
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Liver Cirrhosis; Ascites
Keywords: Cirrhosis; Uncomplicated ascites; Refractory ascites; Chronic albumin treatment
MeSH Terms: conditions — Liver Cirrhosis; Ascites; Fibrosis | interventions — Diuretics; Serum Albumin, Human; Furosemide; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard medical treatment plus albumin (Active Comparator): The patients will receive standard medical treatment (diuretics) plus weekly albumin infusion
  Interventions: Drug: Diuretics plus human albumin
- Standard medical treatment (Other): The patients will receive the standard medical treatment (diuretics), but non albumin for the therapy of ascites
  Interventions: Drug: Diuretics (standard medical treatment)

INTERVENTIONS:
Drug: Diuretics plus human albumin — The patients will receive standard medical treatment plus albumin infusion at the dose of 40 g twice weekly for 2 weeks, and then 40 g weekly for the rest of the study (up to 24 months).
  Other Names: Furosemide and antialdosteronic drugs; Human albumin vials 50 cc 20% solution
  Arms: Standard medical treatment plus albumin
Drug: Diuretics (standard medical treatment) — The patients will receive standard medical treatment (diuretics)
  Other Names: Furosemide and antialdosteronic drugs
  Arms: Standard medical treatment

SUMMARY:
Ascites is the most frequent complication of liver cirrhosis and carries a significant worsening of the prognosis. Approximately 10% of patients per year develop refractory ascites because of either the lack of response to medical treatment or the onset of diuretic-induced complications that preclude the use of an effective dosage. Refractory ascites is associated with an increased incidence of severe complications of cirrhosis. Thus, the overall probability of survival of patients with refractory ascites is very poor, being approximately 30% at 2 years. Repeated large-volume paracentesis, transjugular intrahepatic portosystemic shunt (TIPS), and liver transplantation represent the therapeutic alternatives for refractory ascites. As renal sodium retention and ascites formation are the consequence of portal hypertension and effective hypovolemia, the preservation of the central blood volume represents a major purpose in the management of patients with advanced cirrhosis. Although albumin is responsible for about 70% of the plasma oncotic pressure, the absence of large multicenter randomized studies together with its high cost explains why albumin infusion is not usually included among the therapeutic options for difficult-to-treat ascites.

The objective of the present study is to define the effectiveness of the prolonged administration of human albumin in the treatment of liver cirrhosis with ascitic decompensation. This goal will be reached by performing a multicenter, prospective, randomized clinical trial comparing the efficacy of chronic albumin administration on top of standard medical treatment versus standard medical treatment alone in patients with cirrhosis and ascites.

The study will be conducted in 44 Italian clinical centers and will enrol 440 in- or out-patients affected by liver cirrhosis with uncomplicated ascites who will be randomized with a ratio of 1:1. The duration of the study for each patient is 18 months from randomization. The enrolment of patients will last 18 months and will be competitive between centers. Treatment will be interrupted if one of the following condition occur: orthotopic liver transplantation, TIPS, need of 3 paracentesis/month (indication to TIPS), patient refusal to continue, and medical judgement.

An ancillary optional study will be performed in a subset of patients to analyze the non-oncotic properties of albumin.

DETAILED DESCRIPTION:
Background.

Ascites is the most frequent complication of liver cirrhosis and carries a significant worsening of the prognosis. Medical treatment of uncomplicated ascites is based on diuretics associated to a mild reduction of dietary sodium intake. Approximately 10% of patients per year develop refractory ascites, as defined by the International Ascites Club, because of either the lack of response to medical treatment or the onset of diuretic-induced complications that preclude the use of an effective dosage. Refractory ascites is associated with an increased incidence of severe complications of cirrhosis, such as hepatorenal syndromes (HRS), hyponatremia, spontaneous bacterial peritonitis (SBP), and umbilical hernia rupture and strangulation. Thus, the overall probability of survival of patients with refractory ascites is very poor, being approximately 30% at 2 years. Furthermore, the development of refractory ascites greatly deteriorates the patient's quality of life and substantially raises health costs, due to the frequent need for hospitalization and invasive procedures. Repeated large-volume paracentesis is the most widely accepted therapy for refractory ascites, although early recurrence of fluid accumulation occurs almost invariably. Transjugular intrahepatic portosystemic shunt (TIPS) is usually effective in preventing recurrence, but this procedure can be performed safely only in selected patients. Finally, refractory ascites represents an indication for liver transplantation in patients with no other contraindications.

Renal sodium retention and ascites formation are the consequence of portal hypertension and effective hypovolemia. The background of effective hypovolemia in advanced cirrhosis is represented by arteriolar vasodilation, which mainly occurs in the splanchnic circulatory area and evokes the compensatory activation of neuro-humoral systems able to promote vasoconstriction and renal retention of sodium and water.

Based on the above pathophysiological considerations, the preservation of the central blood volume represents a major purpose in the management of patients with advanced cirrhosis. Albumin constitutes approximately half of the proteins in the plasma of healthy individuals, and is responsible for about 70% of the plasma oncotic pressure. It plays, therefore, a pivotal role in modulating the distribution of fluid between compartments. However, albumin carries other biological properties, such as molecule and drug transport, free radical scavenging, and anti-inflammatory activity, which can be relevant under several circumstances and diseases. Finally, several controlled and/or randomized studies have shown that albumin administration is effective to prevent the circulatory dysfunction after large-volume paracentesis and renal failure after SBP, and to treat HRS when given together with vasoconstrictors. Furthermore, it is currently believed that its capacity to expand central blood volume in cirrhosis is superior to that of several plasma-expanders. In contrast, the chronic use of albumin to treat ascites is still debated, due to the lack of definitive scientific evidence supporting its clinical benefits. Thus, the absence of large multicenter randomized studies together with the high cost of the human albumin explains why albumin infusion is not usually included among the therapeutic options for difficult-to-treat ascites.

Objectives.

The objectives of the present study are to define the effectiveness of the prolonged administration of human albumin in the treatment of liver cirrhosis with ascitic decompensation. This goal will be reached by performing a multicenter, prospective, randomized clinical trial comparing the efficacy of chronic albumin administration on top of standard medical treatment versus standard medical treatment alone in patients with cirrhosis and ascites. The specific objectives of the present study are, therefore, to establish whether or not chronic albumin administration on top of standard medical treatment can improve patient outcomes.

Design of the Study.

The study will be conducted in 42 Italian clinical centers chosen for their high specialization in the management of patients with liver cirrhosis. The study population will consist of 440 in- or out-patients affected by liver cirrhosis with uncomplicated ascites. Patients with cirrhosis and uncomplicated ascites will randomized in two treatment groups:

* standard medical therapy (controls)
* standard medical therapy plus albumin infusion Within 24 hours from randomization, patients will start with albumin infusion at the dose of 40 g twice weekly for 2 weeks, and then 40 g weekly for the rest of the study (up to 18 months). Patients who will develop refractory ascites during the study, will be followed up to completion of the 18 month period or to the need of at least 3 paracentesis/months. Human albumin, as 20% solution - 50 ml, as they are available in the market, will by stored by the hospital Pharmacies of participating Centers and will be given for the patients at the control visits.

Once eligibility to the study will be ascertained, centralized random allocation to the treatment groups will be achieved by means of a web-based service and will be accessible through Internet. Patients will be given an alpha-numeric identification code and randomized in a ratio of 1:1 (standard medical treatment:standard medical treatment plus albumin). Randomization will be stratified according to the following conditions:

* Large volume paracentesis in the last month (yes; no)
* Hyponatremia, as reliable marker of renal function (< 135 mmol/L; ≥ 135 mmol/L) Concomitant Therapies: patients with uncomplicated ascites will be treated with a mild hyposodic diet (approximately 100 mEq/die of Na+) and diuretics. According to the inclusion criteria, patients entering the study will be receiving at least 200 mg/die of an antimineralocorticoid drug and 25 mg/die of furosemide. Dose changes (increase/decrease) of the diuretic therapy will be permitted on the basis on the evolution of ascites decompensation. Total paracentesis can be performed in presence of tense ascites or symptoms due to the accumulation of abdominal fluid and will be followed by the administration of 8 g of albumin per liter of removed ascites. Patients who will develop refractory ascites during the study period will be treated with repeated total paracentesis. TIPS will be considered in patients presenting no other contraindications for this procedure when 3 or more therapeutic paracentesis per month will be needed. Complications such as SBP or HRS will be treated according to current indications, which include albumin infusion. There are any not allowed concomitant medication during the study.

Enrollment: the duration of the study for each patient is 18 months from randomization. The enrollment of patients will last 18 months and will be competitive between centers.

Visit Schedule: after the initial visit, patients will be evaluated every month.

Treatment interruption: each patient is fully entitled to stop his/her participation to the study, at any time. Moreover, patient participation to the study will be interrupted if it will be deemed beneficial to his/her health. Treatment will be interrupted if one of the following condition occur:

* Orthotopic liver transplantation
* TIPS
* Need of 3 paracentesis/month (indication to TIPS)
* Patient refusal to continue
* Medical judgment

Safety Evaluation: the evaluation of human albumin safety will consist in the monitoring and registration of adverse events, serious adverse events, laboratory tests, and vital signs. All events will be managed and reported in compliance with an applicable regulations, and included in the final clinical study report. Specific disease-related adverse events will be collected and documented as part of safety data but will be considered waived from expedited reporting to Regulatory Authorities. In this study, the following SAEs are considered related to the underlying condition and thus will not be considered unexpected unless their course, intensity or other specific features are such that the Investigator, according to his/her best medical judgment, considers these events as exceptional in the context of this medical condition:

* hepatic encephalopathy
* hepatocellular carcinoma
* gastrointestinal bleeding other than variceal bleeding
* bacterial peritonitis
* bacterial infections
* hepatorenal syndrome and renal failure with a non-fatal or fatal outcome
* non-fatal cholestasis
* deterioration of liver function (hyperbilirubinaemia, increased transaminases, coagulopathy)
* serum electrolyte imbalance
* muscle cramps

Statistical Methods.

The study has been designed to demonstrate that the effect of prolonged albumin supplementation improves survival in patients with liver cirrhosis and uncomplicated ascites within 18 months from randomization.

The sample size calculations were based on the primary end-point defined above and calculated by using the Sample Power module included in SPSS11.0, SPSS Inc, Chicago, USA.

- Hypothesis: 35% mortality (due to all causes) in the group of patients undergoing standard medical care and 20% mortality in the group of patients receiving albumin (Wong at al, J Hepatol, 2011). In order to state that the difference in mortality between the two groups is statistically significant with 95% probability, 210 patients per arm have to be enrolled (power 90%). These figures have been calculated assuming a constant drop rate equal to 0.04 per interval.

Ancillary Study.

An ancillary optional study will be performed in a subset of patients to analyze the non-oncotic properties of albumin. This is based on the recent novel observation that the binding, transport, and detoxification capacities of human albumin are severely compromised in patients with liver cirrhosis and this impairment correlates with the degree of liver failure.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of liver cirrhosis (based on clinical, laboratory, endoscopic and ultrasonographic features) and uncomplicated ascites according to the criteria of the International Ascites Club (1).
* Ongoing diuretic treatment with an anti-mineralocorticoid drug at a dose of 200 mg/day and furosemide of 25 mg/day, stable for at least 4 days prior enrollment, not inducing response (defined according to the criteria of the International Ascites Club as body weight reduction ≥ 800 grams in the 4 days prior enrollment). With this limitation, we aim to identify a fairly homogeneous population with a relatively advanced stage of the disease that will likely have more benefit from albumin administration, as also suggested by Gentilini at al. (17).
* Ongoing diuretic treatment with an anti-mineralocorticoid drug at a dose > 200 mg/day and furosemide > 25mg/day, independent of response to treatment.
* EGDS performed in the last 12 months, abdominal ultrasonography performed in the last 30 days, and laboratory tests required by the protocol in the last 7 days.

Exclusion criteria

* Age lower than 18 years
* No written informed consent
* Inability to follow written consent
* Established diagnosis of refractory ascites, as defined by the IAC (1)
* Need of 2 or more paracentesis during the last month
* Serum creatinine > 1.5 mg/dl
* Organic nephropathy, as defined by the IAC (1)
* Hepatorenal syndrome type 1 in the last 15 days
* Gastrointestinal bleeding in the last 15 days
* Ongoing endoscopic eradication after a recent gastro-esophageal variceal bleeding
* Bacterial or fungal infection, including spontaneous bacterial peritonitis, in the last 7 days
* Hepatic encephalopathy grade III/IV
* Budd-Chiari Syndrome
* Patients with TIPS or other surgical porto-caval shunts
* Known and suspected active hepatocellular carcinoma or other malignancies
* Previous liver transplantation
* Ongoing alcohol abuse (patients should be abstinent for at least three months)
* Antiviral therapy for hepatitis B started in the last 6 months
* Heart failure
* Respiratory failure as defined as PO2 <60 mmHg
* Known or suspected hypersensitivity to albumin
* Previous albumin administration given for the treatment of ascites in the last 30 days
* Patients enrolled in other clinical study for the treatment of ascites
* Use of experimental drugs for the last 2 months prior the inclusion in the present study
* Pregnancy and breast-feeding
* Females of child-bearing potential are excluded unless they meet one of the following criteria:

  * Post-menopausal for 6 months or more, and if post-menopausal for less than 2 years, a negative pregnancy test
  * Surgical sterilisation for more than one month duration and a negative pregnancy test
  * Intrauterine device in combination with a secondary barrier (e.g. diaphragm, condom or spermicide) and a negative pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2011-03; Primary Completion 2014-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mortality | 18 months

SECONDARY OUTCOMES:
Incidence of cirrhosis-related clinical complications | 18 months
Number of total paracentesis | 18 months
Number of patients potentially needing TIPS (3 paracentesis/month) | 18 months
Quality of life | 18 months
  QoL will be assessed by the SF-36 and EQ-5D questionnaires
Analysis of the cost/effectiveness ratio | 18 months
Incidence of refractory ascites according to the IAC criteria | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Bernardi, MD, Principal Investigator — University of Bologna; Paolo Caraceni, MD, Study Director — University of Bologna
Locations (33):
- Italy (33):
  - UO Gastroenterology, Riuniti Hospital Of Bergamo, Bergamo, BG
  - UO Internal Medicine, Bentivoglio Hospital, Bologna, Bentivoglio, BO
  - U.O. Semeiotica Medica, Dept. of Clinical Medicine, University of Bologna, Italy, Bologna, BO
  - UO Gastroenterology, General Hospital of Valduce, Como, Como, CO
  - UO Gastroenterology, Hospital of Cosenza, Cosenza, CS
  - Department of Internal Medicine, Bufalini Hospital of Cesena, Cesena, FC
  - UO Gastroenterology, Policlinic Mangiagalli and Regina-Elena of Milan, Milan, MI
  - UO Hepatology and Gastroenterology, Ca' Granda-Niguarda Hospital of Milan, Milan, MI
  - UO Internal Medicine, IRCCS Policlinic S.Donato Milanese, Milan, Milan, MI
  - UO Gastroenterology, University of Modena, Italy, Modena, MO
  - UO Internal Medicine, University of Padova, Padua, PD
  - UO Department of infectious diseases and Hepatology, University of Parma, Parma, PR
  - UO Internal Medicine, Faenza'S Hospital, Italy, Faenza, RA
  - UO Internal Medicine, San Giuseppe Hospital-Marino, Marino, Roma
  - UO Gastroenterology, University of Turine, Torino, TO
  - UO Internal Medicine, University of Udine, Udine, UD
  - UO Internal Medicine, Hospital of Dolo, Venice, Dolo, VE
  - UO Gastroenterology, University of Ancona, Ancona
  - UO Gastroenterology, IRCCS De Bellis, Castellana Grotte-Bari, Bari
  - UO Gastroenterology, University of Bari, Bari
  - UO Internal Medecine, University of Catania, Catania
  - UO Gastroenterology, University of Ferrara, Ferrara
  - UO Internal Medicine, AO University of Florence, Florence
  - UO Internal Medicine, University of Messina, Messina
  - UO Gastroenterology, University of Naples (AO University II), Napoli
  - UO Gastroenterology, University of Naples (Federico II), Napoli
  - UO Internal Medicine, Cotugno Hospital, Naples, Napoli
  - UO Gastroenterology, University of Palermo, Palermo
  - UO Internal Medicine, Hospital Of Rimini, Rimini
  - UO Dept. of Internal Medicine, University of Rome, Policlinic Gemelli Of Rome, Roma
  - UO Gastroenterology, Policlinic Tor Vergata, Rome, Roma
  - UO Gastroenterology, University of Rome, Policlinic Sant'Andrea, Roma
  - UO Gastroenterology, Policlinic Umberto I Rome, Rome

REFERENCES:
- [Background] European Association for the Study of the Liver. EASL clinical practice guidelines on the management of ascites, spontaneous bacterial peritonitis, and hepatorenal syndrome in cirrhosis. J Hepatol. 2010 Sep;53(3):397-417. doi: 10.1016/j.jhep.2010.05.004. Epub 2010 Jun 1. No abstract available. PMID 20633946
- [Background] Runyon BA; AASLD Practice Guidelines Committee. Management of adult patients with ascites due to cirrhosis: an update. Hepatology. 2009 Jun;49(6):2087-107. doi: 10.1002/hep.22853. No abstract available. PMID 19475696
- [Background] Quinlan GJ, Martin GS, Evans TW. Albumin: biochemical properties and therapeutic potential. Hepatology. 2005 Jun;41(6):1211-9. doi: 10.1002/hep.20720. No abstract available. PMID 15915465
- [Background] Gentilini P, Casini-Raggi V, Di Fiore G, Romanelli RG, Buzzelli G, Pinzani M, La Villa G, Laffi G. Albumin improves the response to diuretics in patients with cirrhosis and ascites: results of a randomized, controlled trial. J Hepatol. 1999 Apr;30(4):639-45. doi: 10.1016/s0168-8278(99)80194-9. PMID 10207805
- [Background] Romanelli RG, La Villa G, Barletta G, Vizzutti F, Lanini F, Arena U, Boddi V, Tarquini R, Pantaleo P, Gentilini P, Laffi G. Long-term albumin infusion improves survival in patients with cirrhosis and ascites: an unblinded randomized trial. World J Gastroenterol. 2006 Mar 7;12(9):1403-7. doi: 10.3748/wjg.v12.i9.1403. PMID 16552809
- [Derived] Caraceni P, Riggio O, Angeli P, Alessandria C, Neri S, Foschi FG, Levantesi F, Airoldi A, Boccia S, Svegliati-Baroni G, Fagiuoli S, Romanelli RG, Cozzolongo R, Di Marco V, Sangiovanni V, Morisco F, Toniutto P, Tortora A, De Marco R, Angelico M, Cacciola I, Elia G, Federico A, Massironi S, Guarisco R, Galioto A, Ballardini G, Rendina M, Nardelli S, Piano S, Elia C, Prestianni L, Cappa FM, Cesarini L, Simone L, Pasquale C, Cavallin M, Andrealli A, Fidone F, Ruggeri M, Roncadori A, Baldassarre M, Tufoni M, Zaccherini G, Bernardi M; ANSWER Study Investigators. Long-term albumin administration in decompensated cirrhosis (ANSWER): an open-label randomised trial. Lancet. 2018 Jun 16;391(10138):2417-2429. doi: 10.1016/S0140-6736(18)30840-7. Epub 2018 Jun 1. PMID 29861076
- See also: Official site of the Italian Drug Agency — http://www.agenziafarmaco.it